CLINICAL TRIAL: NCT00753025
Title: Randomized Double Blind Placebo-Controlled Research Of Treatment Efficiency For Patients With Lower Extremity Arteriosclerosis Obliterans By Autologous Transplantation Of Bone Marrow Progenitor Cells
Brief Title: Autologous Bone Marrow For Lower Extremity Ischemia Treating
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinical Center of Cellular Technologies, Russia (Other Government)
Collaborators: Samara State Medical University (Other); Regional hospital of Samara (Unknown)
Responsible Party: Andrey Toropovskiy, Clinical Center of Cellular Technologies, Russia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCCT001
Record Dates: First submitted 2008-09-09; First posted 2008-09-16 (Estimated); Last update posted 2008-09-16 (Estimated); Status verified 2008-09

CONDITIONS: Lower Extremity Ischemia
Keywords: lower extremity ischemia; Bone marrow; Progenitor cells; Neoangiogenesis
MeSH Terms: conditions — Neovascularization, Pathologic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CD133 (Experimental)
  Interventions: Procedure: Bone marrow aspiration , injection of isolated CD 133+ cells
- TNC (Experimental)
  Interventions: Procedure: Bone marrow aspiration, injection of cells
- Placebo (Placebo Comparator)
  Interventions: Procedure: Bone marrow aspiration, injection of saline

INTERVENTIONS:
Procedure: Bone marrow aspiration, injection of cells — Bone marrow is aspirated at patients in all arms.
  Arm "TNC" receives injection of total nucleated cells into ischemic muscle
  Arms: TNC
Procedure: Bone marrow aspiration , injection of isolated CD 133+ cells — arm "CD133" receives injection of isolated CD 133+ cells
  Arms: CD133
Procedure: Bone marrow aspiration, injection of saline — arm "placebo" receives injection of saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether autologous bone marrow derived cells and isolated CD133+ fraction are effective in the treatment limb ischemia

DETAILED DESCRIPTION:
The number of patients with low limb obliterating atherosclerosis steadily grows and compounds more than 20-25 % from all kinds of a cardiovascular pathology. At conservation of this tendency to 2020 the amputation percentage executed due to vessel diseases, can reach 45 %. Hemodynamics improvement in an extremity by surgery is possible at 40 - 70 % of patients even with the widespread and plural lesion of arteries, but results are not always satisfactory. The most actual is the problem of angiosurgical help to patients with distal forms of arterial occlusions, due to the difficulty or impossibility performing reconstructive interventions. In these cases the operations of an indirect revascularization referred on stimulation of a collateral blood flow are carried out. However, despite the reached successes, in some cases results of such interventions do not give desirable effect, search of new methods of treatment therefore is necessary. To date the most perspective methods of neoangiogenesis stimulation are a cellular therapy and gene-engineering technologies. Experimental researches on a model of local limb ischemia showed possibility of use of various cells for neoangiogenesis stimulation. A number of clinical researches at patients with obliterating limb diseases has shown efficacy of cellular therapy even at a critical ischemia. However randomized, the placebo-controlled researches based on principles of evidence based medicine while it is not enough for the convincing conclusions.

ELIGIBILITY:
Inclusion Criteria:

* an obliterating lower extremity atherosclerosis IIB a stage (on Fontaine classification)
* a painless walking distance of 10-50 m
* pulse absence on аа. dorsalis pedis, tibialis posterior, poplitea
* absence of a ischemia in a rest and necrotic changes
* mainly distal form of disease (a lesion of a superficial femoral artery, a popliteal artery, anticnemion arteries) according to an angiography that testifies to impossibility of reconstructive operation performance
* patients after a lumbar sympathectomy and a tibial bone osteoperforations executed previously
* heavy smokers

Exclusion Criteria:

* insulin depended diabetes
* myocardial infarction or a stroke within last year
* an idiopathic hypertensia III stage
* anaemia and other diseases of blood
* decompensation of the chronic diseases which are contraindications to any surgical operation
* HIV infection
* a virus hepatitis
* oncologic diseases
* chemotherapy in the anamnesis

Ages: 39 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-10; Primary Completion 2007-06 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Increasing of painless walking distance | Within the first 30 days, 6 months and 12 months after injection

CONTACTS AND LOCATIONS:
Overall Officials: Olga Tyumina, PhD, Study Director